CLINICAL TRIAL: NCT01804361
Title: Efficacy and Safety Study of Haporine-S in Subjects With Moderate to Severe Dry Eye, A Multicenter, Investigator(Assessor)Blind, Parallel Design, Non-inferiority Phase III Trial
Brief Title: Efficacy and Safety Study of Haporine-S for Treatment of Moderate to Severe Dry Eye Syndromes
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: DH Bio Co., Ltd. (Industry)
Collaborators: BTO Pharm. Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UMT-2012-DH-HS-01; 1360-8040-3073-4190 (Other: Korea Food and Drug Administration)
Record Dates: First submitted 2013-02-27; First posted 2013-03-05 (Estimated); Last update posted 2015-07-22 (Estimated); Status verified 2015-07

CONDITIONS: Dry Eye Syndromes
Keywords: Dry Eye Syndromes
MeSH Terms: conditions — Dry Eye Syndromes | interventions — Cyclosporins

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Haporine-S (Experimental): Moderate to severe dry patients administered with with Haporine-S
  Interventions: Drug: Haporine-S
- Restasis, Cyclosporine 0.05% (Active Comparator): Moderate to severe dry eye patients with Restasis(cyclosporine 0.05%)
  Interventions: Drug: Restasis (cyclosporine 0.05%)

INTERVENTIONS:
Drug: Haporine-S — 1 or 2 drops twice a day at 12 hour interval for 12 weeks
  Arms: Haporine-S
Drug: Restasis (cyclosporine 0.05%) — 1 or 2 drops twice a day at 12 hour interval for 12 weeks
  Arms: Restasis, Cyclosporine 0.05%

SUMMARY:
The purpose of this study is to determine efficacy and safety of Haporine-S eye drop for the patients with moderate to severe dry eye disease in a multicenter phase III clinical trial.

DETAILED DESCRIPTION:
This study is to compare the efficacy and the safety of topical Haposine-S and Restasis® eye drop 0.05% for the patients with moderate to severe dry eye disease in a multicenter, investigator(assessor) blind, parallel design, non-inferiority phase III trial.

Primary outcome is the change of corneal staining score(Oxford scheme) at 12 weeks from baseline.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, age 20 or over
* Patients with moderate to severe dry eye(DEWS Level II or over)
* Be informed of the nature of the study and will give written informed consent

Exclusion Criteria:

* Being treated with steroidal eye drop or non-steroidal anti-inflammatory eye drop for dry eye
* Being treated with systemic steroid or immunosuppressive
* History of eyeball surgical operation within 6 months
* Wearing contact lenses during participation of the study
* Pregnancy or breastfeeding
* Use of cyclosporine eye drop within 2 weeks
* Intraocular pressure(IOP)> 25 mmHg
* History of punctal occlusion within 1 month or during participation of the study
* Hypersensitivity to the investigational products or be suspicious to them
* Patients whom the investigator considers inappropriate to participate in the study

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2013-03; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Corneal staining | up to 12 weeks
  Corneal fluorescein staining will be assessed at 0 day(baseline), 4 weeks and 12 weeks.

SECONDARY OUTCOMES:
Ocular Surface Disease Index(OSID) | 0 day, 4 weeks and 12 weeks
  Ocular Surface Disease Index(OSID) will be assessed at 0 day, 4 weeks and 12 weeks.
Tear Breakup Time(TBUT) | 0 day, 4 weeks and 12 weeks
  Tear Breakup Time(TBUT) will be assessed at 0 day(baseline), 4 weeks and 12 weeks.
Schirmer score | 0 day, 4 weeks and 12 weeks
  Schirmer score will be assessed at 0 day(baseline), 4 weeks and 12 weeks.
Drug compliance | 0 day, 4 weeks and 12 weeks
  Drug compliance(conjunctival hyperemia and burning etc) will be assessed at 0 day(baseline), 4 weeks and 12 weeks.
DEWS(Dry Eye WorkShop) level | 0 day, 4 weeks and 12 weeks
  Level on dry eye severity grading scheme of DEWS will be assessed at 0 day(baseline), 4 weeks and 12 weeks.

OTHER OUTCOMES:
Adverse Events | 1 year
  Adverse Event will be assessed for the whole study period(1 year).
Serious Adverse Events | 1 year
  Serious Adverse Event will be assessed for the whole study period(1 year).

CONTACTS AND LOCATIONS:
Overall Officials: Hyo-Myung KIM, MD, PhD, Principal Investigator — Korea University Anam Hospital; Jong Suk SONG, MD, PhD, Principal Investigator — Korea University Guro Hospital; Hyung Keun LEE, MD, PhD, Principal Investigator — Yonsei University Gangnam Severance Hospital; Jong-Soo LEE, MD, PhD, Principal Investigator — Busan National University Hospital; Mee Kum KIM, MD, PhD, Principal Investigator — Seoul National University Hospital; Myoung-Joon KIM, MD, PhD, Principal Investigator — Asan Medical Center
Locations (6):
- South Korea (6):
  - Busan National University Hospital, Busan, Busan
  - Seoul National University Hospital, Seoul, Seoul
  - Yonsei University Gangnam Severance Hospital, Seoul, Seoul
  - Korea University Anam Hospital, Seoul, Seoul
  - Asan Medical Center, Seoul, Seoul
  - Korea University Guro Hospital, Seoul, Seoul